# Comparison of Biologicals in Treatment of Severe Asthma (BiSA)

NCT04158050

Reviewed and accepted by the Hospital Research Board 2<sup>nd</sup> Jan 2018 and 4<sup>th</sup> Sept 2019 (HUS/64/2018 and HUS/25/2019)

Astman hoitotulokset Suomessa – biologiset lääkkeet, digihoitopolku ja iäkkäät Asthma treatment results in Finland – biologicals, digital health pathway and elderly patients

### Lyhennelmä

Astman hoitotulokset on tutkimus, jossa selvitetään biologisista lääkkeistä saatavaa hyötyä tavanomaiseen kliiniseen potilasmateriaaliin sekä digihoitopolun käyttökelpoisuutta astman hoidossa sekä iäkkäiden astmaa sairastavien erityispiirteitä.

- 1) Ensimmäisen osatyön tavoitteena oli selvittää, ovatko **astman biologisia lääkehoitoja saaneet astmapotilaat hyötyneet lääkityksestä** (tutkittavien lukumäärä noin 60).
- 2) Toisen osatyön tavoitteena on selvittää, astman biologisia lääkehoitoja saaneiden potilaiden tilanne ja hoitovaste ylähengitystiesairauden (krooninen rinosinuiitti) osalta sekä keuhkojen kuvantamislöydökset (tutkittavien lukumäärä noin 60) (ovatko ylähengitystieoireet ja löydökset vähentyneet biol. lääkkeiden myötä ja korreloivatko HRCT-löydökset ysköslöydöksiin)
- 3) Kolmannen osatyön tavoitteena on arvioida astman **digihoitopolun vaikutuksia astman hoitotuloksiin** (100 potilasta).
- 4) Neljännessä osatyössä tavoitteena on arvioida astman hoitotuloksia astman laaturekisterin näkökulmasta 2 vuoden seurannassa erityisesti iäkkäiden 65-vuotiaiden hoitoa koskien. Hoitotuloksia arvioidaan suhteessa erilaisiin ilmiasuihin pahenemisvaiheiden, keuhkojen toimintakokeiden tulosten, oireiden ja lääkityksen tarpeen perusteella (100 potilasta).

#### Abridgment

Asthma treatment results is a study that investigates the benefit of biological drugs to conventional clinical patient material, as well as the usefulness of the digital treatment path in the treatment of asthma, as well as the special characteristics of elderly people with asthma.

- 1) The aim of the first part of the work was to find out whether asthma patients who received biological drug treatments for asthma have benefited from the medication (number of subjects approximately 60).
- 2) The aim of the second part of the work is to find out the situation and treatment response of patients who have received biological drug treatments for asthma with regard to upper respiratory disease (chronic rhinosinusitis) and lung imaging findings (number of subjects about 60) (whether upper respiratory symptoms and findings have decreased with biological drugs and whether HRCT findings correlate with sputum findings)
- 3) The goal of the third part of the work is to evaluate the effects of the digital asthma treatment path on asthma treatment results (100 patients).
- 4) In the fourth part, the goal is to evaluate the results of asthma treatment from the perspective of the asthma quality register in a 2-year follow-up, especially regarding the treatment of elderly people aged 65 years. Treatment results are evaluated in relation to various manifestations based on exacerbations, lung function test results, symptoms and the need for medication (100 patients).

#### Johdanto

Astma on pitkäaikainen keuhkosairaus, johon liittyy keuhkoputkien inflammaatio ja niiden supistumisherkkyys. Suomessa astmaa sairastaa 9% väestöstä, ja arvioiden mukaan esiintyvyys on viime vuosikymmenien aikana lisääntynyt. Vaikeaa astmaa sairastaa kansainvälisten tutkimusten mukaan 3-10% kaikista astmaatikoista, ja tähän potilasryhmään kuluu merkittävä osa astmaan käytetyistä terveydenhuollon resursseista. (Harju, T 2012)

European Respiratory Society:n (ERS) mukaan vaikea astma määritellään astmana, joka edellisen vuoden aikana on vaatinut suuriannoksista inhalaatiosteroidia sekä lisäksi pitkävaikutteista beetaagonistia, leukotrieenireseptorisaplaajaa, teofylliiniä ja/tai jatkuvaa tai lähes jatkuvaa systeemisesti annosteltua steroidia pysyäkseen tasapainossa (Chung 2014). Vaikeaksi määritellään myös astma, joka ei ylläolevista hoidoista huolimatta pysy tasapainossa. Epätasapainossa olevaa astmaa kuvaa jatkuva oireilu, toistuvat pahenemisvaiheet, vakavat sairaalahoitoon, tehohoitoon tai mekaaniseen ventilaatioon johtaneet pahenemisvaiheet sekä keuhkofunktion alenema FEV1:llä mitattuna.

Vaikean astman on tutkimuksissa havaittu olevan hyvin heterogeeninen tila, jossa taudin ilmentyminen ja vaste perinteisille astman lääkehoidoille eri henkilöillä vaihtelee (McCracken JL 2017). Niin kutsuttu astman fenotyypitys on viime vuosina herättänyt tutkijoiden mielenkiinnon, tavoitteena on löytää astman eri fenotyypeille spesifejä biomarkkereita astman uusien lääkehoitojen kohdemolekyyleiksi.

#### Astman erilaiset ilmiasut ja tulehdukselliset alamuodot

Tutkimuksissa on havaittu astman fenotyyppejä, joihin liittyy vaihtelevissa määrin esimerkiksi eosinofiliaa, atopiaa ja lihavuutta (Fajt 2015). Eri fenotyypeissä inflammaation ja oireiden osuus sekä keuhkofunktiot vaihtelevat. Toistuvat pahenemisvaiheet ovat tavallisempia vaikeassa astmassa ylipainoisilla ja tupakoivilla henkilöillä. Vaikeaan astmaan liittyy usein samaan aikaan esiintyviä muita sairauksia ja tiloja, jotka huonontavat osaltaan astman tasapainoa tai jotka on huomioitava erotusdiagnostisina tekijöinä hengenahdistuksen osalta (McCracken JL 2017, Papi 2018). Tällaisia tiloja ovat esim. refluksitauti, nenäpolyypit ja rinosinuiitti, toiminnallinen äänihuulisalpaus, lihavuus, obstruktiivinen uniapnea, hyperventilaatiosyndrooma, tupakointi tai siihen liittyvä sairaus, psyykkiset tekijät, hormonaaliset tekijät ja lääkeaineet (tulehduskipulääkkeet, aspiriini, beetasalpaajat, ACE-estäjät) (Wechsler ME, 2014).

Vaikeassa astmassa inflammaatiota voi dominoida eosinofiilit tai neutrofiilit, tai vaihtoehtoisesti tulehduksessa vaikuttavat rinnakkain sekä neutrofiilit että eosinofiilit, tai ei kumpikaan. Tulehdussolujen määrää ja jakaumaa on tutkittu sylkinäytteistä, bronkoalveolaarisista lavaationäytteistä ja keuhkoputkista otetuista koepaloista. Vaikeimmat astman ilmentymät ovat assosioituneet tulehdukseen, jossa on sekä neutrofiileja että eosinofiileja.

Eosinofiilisessä tulehduksessa keskeisenä on tyypin 2 inflammaatiovaste, jossa Th2-auttajasoluista peräisin olevat sytokiinit (interleukiini-4, -5 ja -13) edistävät immunoglobuliini E:n (IgE) eritystä plasmasoluista ja mm. eosinofiilien migraatiota ja aktivaatiota. Eosinofiilit puolestaan erittävät sytokiineja, jotka edistävät tulehdusta ja sitä kautta hengitysteiden dysfunktiota. Th2-tulehdusvasteen voi indusoida esimerkiksi allergeeni, infektio tai jokin ulkoinen ärsyke. Eosinofiilisen vaikean astman patogeneesissa tärkeä välittäjäaine on myös interleukiini-5 (IL-5), joka myötävaikuttaa eosinofiilien erilaistumiseen, migraatioon ja aktivaatioon. IL-5 on sytokiini, jota erittävät ainakin lymfosyytit ja syöttösolut, mutta mahdollisesti myös eosinofiilit itse. Neutrofiilisen tulehduksen mekanismit vaikeassa astmassa ovat edelleen puutteellisesti tunnettuja. Osalla vaikeaa astmaa sairastavista hengitysteissä ei kuitenkaan enää näy merkkejä kummastakaan ylläolevasta tulehdusprosessista, jolloin on käytetty nimitystä "paucigranulocytic asthma". Myös tässä ryhmässä vaikean astman mekanismit ovat vielä epäselvät ja vaativat lisätutkimuksia. (Darveaux J, 2016, Israel E, 2017)

### Vaikean astman biologiset lääkkeet

Yllä kuvattuja vaikean astman tulehdusmekanismeja on hyödynnetty uusien, kohdennettujen biologisten lääkkeiden kehittämisessä. Tällä hetkellä Suomessa on käytössä IgE-vasta-aine omalitsumabi vaikeassa allergisessa astmassa ja IL-5 vasta-aineet mepolitsumabi ja reslitsumabi vaikeassa eosinofiilisessa astmassa (Boyman O). Biologisten lääkkeiden hyödyistä vaikean astman hoidossa tarvitaan vielä lisätutkimuksia, ja erityisesti potilaiden valikoimisessa biologiseen lääkehoitoon tarvitaan lisää tietoa ja kokemusta.

Omalitsumabi on monoklonaalinen IgE-vasta-aine, joka estää IgE:n sitoutumisen sen reseptoriin syöttösoluissa, dendriittisoluissa, basofiileissa, eosinofiileissa ja Langerhansin soluissa. Omalitsumabi on ensimmäinen vaikean allergisen astman hoitoon hyväksytty monoklonaalinen vasta-aine. (Normansell R 2014). Selvin näyttö on nähty pahenemisvaiheiden vähenemisessä. Mepolitsumabi on monoklonaalinen IL-5-vasta-aine, jonka vaikutus vaikeassa eosinofiilisessa astmassa kohdistuu eosinofiilisen tulehduksen vähentämiseen. Mepolitsumabin on tutkimuksissa

ositettu vähentävän pahenemisvaiheita vaikeassa eosinofiilisessä astmassa, ja se vaikuttaa myös parantavan elämänlaatua ja vähentävän syljen ja veren eosinofiilitasoja (Liu Y 2013). Reslitsumabi on humanisoitu IgG4-kappa monoklonaalinen IL-5-vasta-aine, jota käytetään vaikean eosinofiilisen astman hoidossa, kun muu lääkitys on riittämätön. (Castro, M)

### Astman digihoitopolku ja astmarekisteri

Helsingin ja Uudenmaan sairaanhoitopiirissä on käytössä astman digihoitopolku, joka toimii erikoissairaanhoidon täydentävänä työkaluna. Digihoitopolku tarjoaa yhteydenottokanavan hoitavaan yksikköön vistien tai etävastaanottojen kautta, työkaluja oireiden ja terveysarvojen seurantaan, potilasohjeita ja omahoito-ohjelmia. Digihoitopolun kautta voidaan myös siirtää potilaan laitetietoja terveydenhuollon henkilökunnalle nähtäviksi. Digihoitopolun käyttö on maksutonta mutta vaatii hoitosuhteen hoitavaan yksikköön. Digihoitopolun avulla voidaan lisätä potilaan omaa osallistumista hoitoon ja parantaa tiedonkulkua potilaan ja hoitava yksikön välillä. Astman digihoitopolun vaikuttavauutta erikoissairaanhoidossa hoidettujen astmapotilaiden hoitotuloksiin ei ole vielä systemaattisesti analysoitu.

Astmarekisteri on toukokuussa 2018 käyttöön otettu sähköinen alusta astmapotilaiden hoidon seurantaan. Kyseessä on yksi valtakunnallisessa käytössä olevista BCBMedicalin rakentamista ja ylläpitämistä laaturekistereistä, joita kaikkiaan eri sairauksiin on Suomessa käytössä yli 70. Kyseessä on järjestelmä, jonka tarkoituksena on tuottaa astmapotilaiden sairauden vaikeusasteesta ja hoidon laadusta helposti kerättävää, käytettävää, vertailtavaa ja raportoitavaa tietoa. Astmarekisteri käyttää osin hyödykseen sähköisen sairauskertomusjärjestelmän diagnoosi-, lääke- ja laboratoriotulostietoja ja osin hoidon myötä kertyvää tietoa tallennetaan astmapotilaan käyntien yhteydessä rekisteriin.

### 2. Tavoitteet

Tavoitteena on väitöskirja, joka tulee koostumaan kolmesta osatyöstä. Ensimmäinen osatyö arvioitavana

- 1) Ensimmäisen osatyön tavoitteena oli selvittää, ovatko **astman biologisia lääkehoitoja saaneet astmapotilaat hyötyneet lääkityksestä pahenemisvaiheiden vähentymisenä**, tablettikortisonin tai mikrobilääkekuurien käytön vähenemisenä, astmaoireiden vähenemisenä tai keuhkojen toimintakokeiden tulosten paranemisena.
- 2) Toisen osatyön tavoitteena on selvittää, astman biologisia lääkehoitoja saaneiden potilaiden tilanne ja hoitovaste ylähengitystiesairauden (krooninen rinosinuiitti) osalta sekä keuhkojen kuvantamislöydökset (HRCT: atelektaasi, bronkiektasiat, bronkusten paksuseinäisyys, nodulukset, limatulpat, mattalasimuutokset, ilmasalpaus, retikulaatiota (0 ei lainkaan, 1 toisella puolella, 2 molemmilla puolilla).

Täydennetään tiedot uusien hoitoja aloittaneiden osalta ja muiltakin tarpeen mukaan: ikä, sp, tupakointi (askivuodet), krooninen/allerginen nuha, osteoporoosi, em HRCT-löydökset, BMI, OCS ennen biologisia hoitoja ja viimeisin tieto, OCS kuurit 12 kk aikana ja viimeisin tieto, päivystyskäynnit, antibioottihoidot, B-eos ennen ja viimeisin, ACT ennen hoitoa ja viimeisin, FEV1 (l, %, Z), FVC (l, %, Z), FEV1/FVC (l, %, Z), S-IgE, prick-positiivisuus (kissa, koira, koivu, timotei, pölypunkki, Aspergillus fumigatus), liitännäissairaudet (MCC, HTA, refluksi, osteoporoosi, COPD, flimmeri, uniapnea, DM, hypotyreoosi, masennus, ahdistuneisuushäiriö), yskösten bakteeri-, sieni- ja mykobakteeriviljelynäytetulokset (viimeisimmät jos otettu useita, mikrobin nimi, +/++/+++). Täydennetään tietoihin: inhalaatiosteroidi (vrk-annos), po steroidi (vrk-annos), LABA, LAMA, SABA, montelukasti, teofylliini (kyllä/ei).

Ylähengitystielöydösten osalta arvioidaan seuraavia: NSO: nestevaakapinnat, limakalvoturvotus, polyypit; krooninen rinosinuiitti 0 = ei, 1 = kyllä (KNK- tai keuhkolääkärin arvio), allerginen nuha 0/1. FESS, pelkkä polyyppien poisto eli polypektomia, etmoidektomia; antibioottikuuri(t) sinuiittiin status: nenäpolypoosia (0/1) tai märkää KNK-statuksessa; nenästeroidi kyllä/ei, montelukasti kyllä/ei, po steroidi jatkuvana tai kuureina (annos); punktion viljelylöydös (viimeisimmät jos otettu useita, mikrobin nimi, +/++/+++). Lisäksi merkitään biologinen lääkehoito, aloitettu (päivä), kuinka kauan käytetty (kuukausina), ylähengitystieoireiden ilmeneminen biol lääkkeiden aloituksen jälkeen (pahentunut, ennallaan, parantunut), ovatko polyypit uusituneet tai pahentuneet, onko ylähengitystietoimenpiteitä tehty biologisten lääkkeiden aloitusten jälkeen.

- 3) Kolmannen osatyön tavoitteena on arvioida astman **digihoitopolun vaikutuksia astman hoitotuloksiin**. Tavoitteena on verrata astman digihoitopolun mukaisesti hoidettujen astmapotilaiden pahenemisvaiheiden määrää, oireita, keuhkojen toimintakokeiden tuloksia ja lääkityksen tarvetta astmapotilaisiin, joita ei ole hoidettu hoitopolulla.
- 4) Neljännessä osatyössä tavoitteena on arvioida astman hoitotuloksia astman laaturekisterin näkökulmasta 2 vuoden seurannassa erityisesti iäkkäiden 65-vuotiaiden hoitoa koskien. Hoitotuloksia arvioidaan suhteessa erilaisiin ilmiasuihin pahenemisvaiheiden, keuhkojen toimintakokeiden tulosten, oireiden ja lääkityksen tarpeen perusteella.

#### 3. Suunnitelma

Ensimmäiseen osatyöhön haettiin tiedot sairaskertomusmerkinnöistä vaikeaa astmaa sairastavista ja HUS-alueella biologisia lääkehoitoja saaneista 2009 lähtien. Kyseessä oli takautuva tutkimus. Toisessa osatyössä haetaan tiedot n. 50 potilaasta, joita on hoidettu astman digipolulla, ja 50 potilaasta, joita vastaavaan aikaan tavanomaisesti ei-digihoitopolkua hyödyntäen, on hoidettu Iho- ja allergiasairaalan allergiayksikössä (HGD Study, HUH Goes Digital Study). Haettavia tietoja ovat pahenemisvaiheet, oireet astman oirekyselyllä arvioituna, keuhkojen toimintakokeiden tulokset ja lääkityksen tarve. Tietojen perusteella arvioidaan, onko ryhmien välillä eroa hoitotasapainossa 1 ja 2 vuoden seurantaajan jälkeen. Kolmannessa osatyössä hyödynnetään tällä hetkellä n. 1500 18-vuotiaan tai sitä vanhemman potilaan kattavaa astman laaturekisteriä ja arvioidaan astman hoitotuloksia erityisesti yli 65-vuotiaiden ikäryhmässä (n = 250) pahenemisvaiheiden, oireiden, keuhkojen toimintakokeiden tulosten ja lääkityksen tarpeen perusteella 2 vuoden seurannassa.

### 4. Aikataulu ja kustannusarvio

Potilastietojen keruu ja tulosten analysointi tehdään toisen osatyön osalta vuoden 2019 ja kevään 2020 aikana, ja kolmannen osatyön osalta vuosien 2020 ja 2021 aikana. Väitöskirjan kirjoittaminen ja tohtorikoulutukseen kuuluvien opintojen suorittaminen suunnitellaan tehtäväksi vuoteen 2023 mennessä. Kustannusarvio osatöiden toteuttamiselle vuosien 2019-20 aikana 2 kuukauden tutkimusvapaan muodossa on 5000 euroa (2500 euroa/kk).

## 5. Tulosten merkitys ja hyödynnettävyys

Ensimmäisen osatyön tuloksia hyödynnetään arvioimalla HUS-alueen vaikeaa astmaa sairastavien tarvetta ja hyötyä astman biologisiin lääkkeisiin liittyen. Tuloksia voidaan käyttää suoraan omaa

toimintaa ohjaavana. Toisen ja kolmannen osatyön tuloksia hyödynnetään astman hoitoketjujen kehittämiseen, astman hoidon laadun arvioimiseen Suomessa ja hoitomuotojen kehittämiseen.

# 6. Tutkimusryhmä

Emma Kotisalmi, LL, keuhkosairauksiin ja allergologiaan erikoistuva lääkäri, HUS sydänkeuhkokeskus Meilahden ja Jorvin sairaala

Paula Kauppi, dos, oyl, keuhkosairauksien ja allergologian el, IAS

Witold Mazur, dos. oyl, keuhkosairauksien ja allergologian el, HUS Sydän- ja keuhkokeskus

Mika Mäkelä, dos., lastentautien ja lastenallergologian erikoislääkäri, professori, IAS

Auli Hakulinen, LL, keuhkosairauksien erikoislääkäri, IAS

Hilkka Viitanen, LL, keuhkosairauksien ja allergologian el, IAS

Timo Helin, LL, sisätautien sekä keuhkosairauksien ja allergologian erikoislääkäri, IAS

Tuuli Thomander, LK, Itä-Suomen yliopisto

# 7. Kirjallisuusviitteet

- 1. Chung KF, Wenzel SE, Brozek JL, Bush A, Castro M, Sterk PJ, Adcock IM, Bateman ED, Bel EH, Bleecker ER, Boulet LP, Brightling C, Chanez P, Dahlen SE, Djuckanovic R, Frey U, Gaga M, Gibson P, Hamid Q, Jajour NN, Mauad T, Sorkness RL, Teague WG. International ERS/ATS guidelines on definition, evaluation and treatment of severe asthma. Eur Respir J2014; 43: 343-373.
- 2. McCracken JL, Veeranki SP, Ameredes PT, Calhoun JC. Diagnosis and management of asthma in adults, a review. JAMA 2017; 318: 279-290.
- 3. Fajt M, Wenzel SE. Asthma phenotypes and the use of biologic medications in asthma and allergic disease: the next steps toward personalized care. J Allergy Clin Immunol 2015; 135: 299-310.
- 4. Papi A, Brightling C, Pedersen SE, Reddel HK. Asthma. Lancet 2018; 391(10122):783-800. doi: 10.1016/S0140-6736(17)33311-1.
- 5. Israel E, Reddel HK. Severe and Difficult-to-Treat Asthma in Adults. N Engl J Med 2017; 377: 965-76.
- 6. Darveaux J, Busse WW. Biologics in asthma--the next step toward personalized treatment. J Allergy Clin Immunol Pract 2015 Mar-Apr;3(2):152-60; quiz 161. doi: 10.1016/j.jaip.2014.09.014.
- 7. Boyman O, Kaegi C, Akdis M, Bavbek S, Bossios A, Chatzipetrou A, Eiwegger T, Firinu D, Harr T, Knol E, Matucci A, Palomares O, Schmidt-Weber C, Simon HU, Steiner UC, Vultaggio A, Akdis CA, Spertini F. EAACI IG Biologicals task force paper on the use of biological agents in allergic disorders. Allergy 2015; 70: 727-754.
- 8. Normansell R, Walker S, Milan SJ, Walters EH, Nair P. <u>Omalizumab for asthma in adults and children.</u> Cochrane Database Syst Rev. 2014 Jan 13;(1):CD003559. doi: 10.1002/14651858.CD003559.pub4. Review.
- 9. Patel TR, Sur S. IgE and eosinophils as therapeutic targets in asthma. Curr Opin Allergy Clin Immunol 2017 Feb;17(1):42-49. doi: 10.1097/ACI.00000000000336.

- 10. Walker S, Monteil M, Phelan K, Lasserson TJ, Walters EH. <u>Anti-IgE for chronic asthma in adults and children.</u> Cochrane Database Syst Rev. 2006 Apr 19;(2):CD003559. Review. Update in: Cochrane Database Syst Rev. 2014;1:CD003559.
- 11. Liu Y, Zhang S, Li DW, Jiang SJ. Efficacy of anti-interleukin-5 therapy with mepolizumab in patients with asthma: a meta-analysis of randomized placebo-controlled trials. PLoS One 2013; 8:e59872.
- 12. Katial RK, Bensch GW, Busse WW, et al. Changing Paradigms in the Treatment of Severe Asthma: The Role of Biologic Therapies. J Allergy Clin Immunol Pract 2017;5(2S):S1-S14. doi: 10.1016/j.jaip.2016.11.029.
- 13. <u>Castro M</u>, <u>Mathur S</u>, <u>Hargreave F</u> ym. <u>Am J Respir Crit Care Med.</u> Reslizumab for poorly controlled, eosinophilic asthma: a randomized, placebo-controlled study. 2011;184:1125-32.
- 14. Cabon Y, Molinari N, Marin G, Vachier I, Gamez AS, Chanez P, Bourdin A. A comparison of anti-interleukin-5 therapies in patients with severe asthma: a global and indirect meta-analyses of randomized placebo-controlled trials. Clin Exp Allergy. 2017 Jan;47(1):129-138. doi: 10.1111/cea.12853. Epub 2016 Dec 8. Review.
- 15. Cockle SM, Stynes G, Gunsoy NB, Parks D, Alfonso-Cristancho R, Wex J, Bradford ES, Albers FC, Willson J. <u>Comparative effectiveness of mepolizumab and omalizumab in severe asthma: An indirect treatment comparison.</u> Respir Med. 2017 Feb;123:140-148. doi: 10.1016/j.rmed.2016.12.009.
- 16. Chupp GL, Bradford ES, Albers FC, Bratton DJ, Wang-Jairaj J, Nelsen LM, Trevor JL, Magnan A, Ten Brinke A. Efficacy of mepolizumab add-on therapy on health-related quality of life and markers of asthma control in severe eosinophilic asthma (MUSCA): a randomised, double-blind, placebo-controlled, parallel-group, multicentre, phase 3b trial. Lancet Respir Med. 2017 May;5(5):390-400. doi: 10.1016/S2213-2600(17)30125-X.
- 17. Farne HA, Wilson A, Powell C, Bax L, Milan SJ. <u>Anti-IL5 therapies for asthma.</u> Cochrane Database Syst Rev. 2017 Sep 21;9:CD010834. doi: 10.1002/14651858.CD010834.pub3. Review.
- 18. Humbert M, Taillé C, Mala L, Le Gros V, Just J, Molimard M; STELLAIR investigators. Omalizumab effectiveness in patients with severe allergic asthma according to blood eosinophil count: the STELLAIR study. Eur Respir J. 2018 May 10;51(5). pii: 1702523. doi: 10.1183/13993003.02523-2017. Print 2018 May.
- 19. Maselli DJ, Velez MI, Rogers L. Reslizumab in the management of poorly controlled asthma: the data so far. J Asthma Allergy. 2016 Aug 31;9:155-62. doi: 10.2147/JAA.S94164. eCollection 2016. Review
- 20. Castillo JR, Peters SP, Busse WW. Asthma Exacerbations: Pathogenesis, Prevention, and Treatment. J Allergy Clin Immunol Pract. 2017 Jul Aug;5(4):918-927. doi: 10.1016/j.jaip.2017.05.001. Review.
- 21. Sabogal Piñeros YS, Bal SM, van de Pol MA, Dierdorp BS, Dekker T, Dijkhuis A, Brinkman P, van der Sluijs KF, Zwinderman AH, Majoor CJ, Bonta PI, Ravanetti L, Sterk PJ, Lutter R. Anti-IL5 in mild asthma alters rhinovirus-induced macrophage, B cell and neutrophil responses (MATERIAL): a placebo-controlled, double-blind study. Am J Respir Crit Care Med. 2018 Sep 7. doi: 10.1164/rccm.201803-0461OC. [Epub ahead of print]

- 22. <u>Caminati M, Pham DL</u>, <u>Bagnasco D</u>, <u>Canonica GW</u>. Type 2 immunity in asthma. World Allergy Organ J 2018: 11(1): 13. doi: 10.1186/s40413-018-0192-5. eCollection 2018.
- 23. Panettieri RA Jr, Sjöbring U, Péterffy A, Wessman P, Bowen K, Piper E, Colice G, Brightling CE. <u>Tralokinumab for severe, uncontrolled asthma (STRATOS 1 and STRATOS 2): two randomised, double-blind, placebo-controlled, phase 3 clinical trials.</u> Lancet Respir Med. 2018 Jul;6(7):511-525. doi: 10.1016/S2213-2600(18)30184-X.
- 24. <a href="https://www.terveyskylä.fi/allergia-astmatalo">https://www.terveyskylä.fi/allergia-astmatalo</a>.
- 25. https://www.terveyskirjasto.fi
- 26. Bonini M, Usmani OS. Novel methods for device and adherence monitoring in asthma. Curr Opin Pulm Med 2018; 24: 63-69.
- 27. Merivuori T, Tapanainen H. Astma avoterveydenhuollossa, Duodecim 2019.
- 28. Tsiligianni I, Goodridge D, Marciniuk D, Hull S, Bourbeau J. Four patients with a history of acute exacerbations of COPD: implementing the CHEST/Canadian Thoracic Society guidelines for preventing exacerbations. NPJ Prim Care Respir Med. 2015 May 7;25:15023. doi: 10.1038/npjpcrm.2015.23.
- 29. Ambrosino N, Makhabah DN, Sutanto YS. Tele-medicine in respiratory diseases. Multidiscip Respir Med. 2017 Apr 20;12:9. doi: 10.1186/s40248-017-0090-7. eCollection 2017. Review.
- 30. Huang X, Matricardi PM. Allergy and asthma care in the mobile phone era. Clin Rev Allergy Immunol. 2016 May 21. [Epub ahead of print] Review.
- 31. Lombardi C, Bonini M, Passalacqua G. Mobile Apps Multicenter Italian Study Group. Eur Ann Allergy Clin Immunol 2018; 50: 268-272.
- 32. Morton K, Dennison L, May C, Murray E, Little P, McManus RJ, Yardley L. Using digital interventions for self-manament of chronic physical health conditions: a metaethnography review of published studies. Patient Educ Couns. 2017 Apr;100(4):616-635. doi: 10.1016/j.pec.2016.10.019. Epub 2016 Oct 20. Review.

Taulukko 1. Alustava arvio biologisia lääkehoitoja saaneiden potilaiden taustamuuttujista.

| Characteristics | Reslizumab, | Mepolizumab, n=13 | Omalizumab, n=24 | Infliximab, n=1 |
|---|---|---|---|---|
| | n=11 | | | |
| Time of use (months) | 5.50 (1-12. SD | 8.77 (1-16. SD 4.99) | 38.22 (1-109. SD | 70 |
| | 3.20) | | 31.87) | |
| Age (years) | 55 (37-70. SD | 57 (30-71. SD 10.12) | 47 (27-74. SD 10.69) | 47 |
| | 9.96) | | | |
| Women (number, (%)) | 5 (45) | 8 (62) | 17 (71) | 1 (100) |
| Smokers (number, (%)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) |
| Ex-smokers (number, | 5 (45) | 4 (31) | 3 (13) | 0 (0) |
| (%)) | ` ′ | | , , | . , |
| Nasal polyposis | 10 (91) | 8 (62) | 13 (54) | 0 (0) |
| (number, (%)) | | | | |
| Chronic/allergic rhinitis | 9 (82) | 11 (85) | 24 (100) | 0 (0) |
| (number, (%)) | , í | , , | , , | |
| Positive skin prick test | 3 (27) | 4 (31) | 19 (79) | 1 (100) |
| (number, (%)) | , , | | | , , |
| HRCT findings * | 9 (82) | 10 (77) | 14 (58) | 0 (0) |
| (number, (%)) | , í | , , | | ` ' |
| Mean daily OCS dose | 9.04 (0-20. SD | 10.58 (0-40. SD | 4.42 (0-20. SD 6.37) | 16 |
| before treatment ** | 4.87) | 9.31) | | |
| (mg) | · | | | |
| FEV1 before treatment | 2.72 (SD 0.85) | 2.14 (SD 0.64) | 2.75 (SD 0.87) | 2.62 |
| (liters) | | | | |
| FVC before treatment | 3.87 (SD 1.05) | 3.20 (SD 0.93) | 3.72 (SD 0.87) | 3.28 |
| (liters) | ĺ | | , , , , , | |
| FEV1/FVC before | 0.70 (SD 0.10) | 0.68 (SD 0.13) | 0.74 (SD 0.13) | 0.80 |
| treatment | | | | |
| Blood eosinophil count | 0.51 (SD 0.49) | 0.46 (SD 0.38) | 0.42 (SD 0.39) | 0 |
| before treatment | | | | |
| (E9/liter) | | | | |

#### Introduction

Asthma is a long-term lung disease that involves inflammation of the bronchial tubes and their sensitivity to contraction. In Finland, 9% of the population suffers from asthma, and according to estimates, the prevalence has increased in recent decades. According to international studies, 3-10% of all asthmatics suffer from severe asthma, and this group of patients consumes a significant part of the health care resources used for asthma. (Harju, T 2012) According to the European Respiratory Society (ERS), severe asthma is defined as asthma that, during the previous year, has required high-dose inhaled steroid plus a long-acting beta-agonist, leukotriene receptor blocker, theophylline and/or continuous or near-continuous systemically dosed steroid to maintain balance (Chung 2014). Asthma that does not remain balanced despite the above treatments is also defined as severe. Unbalanced asthma is characterized by persistent symptoms, frequent exacerbations, severe exacerbations leading to hospitalization, intensive care or mechanical ventilation, and decreased lung function as measured by FEV1. Severe asthma has been found in studies to be a very heterogeneous condition, in which the manifestation of the disease and the response to traditional asthma medical treatments in different individuals varies (McCracken JL 2017). The so-called asthma phenotyping has attracted the interest of researchers in recent years, the goal is to find specific biomarkers for different asthma

The different manifestations and inflammatory subtypes of asthma

phenotypes as target molecules for new asthma drug treatments.

Asthma phenotypes have been observed in studies, which are associated to varying degrees with, for example, eosinophilia, atopy and obesity (Fajt 2015). In different phenotypes, the proportion of inflammation and symptoms and lung functions vary. Repeated exacerbations are more common in severe asthma in people who are overweight and who smoke. Severe asthma is often associated with other diseases and conditions occurring at the same time, which contribute to worsening the

balance of asthma or which must be taken into account as differential diagnostic factors for shortness of breath (McCracken JL 2017, Papi 2018). Such conditions include e.g. reflux disease, nasal polyps and rhinosinusitis, functional vocal cord obstruction, obesity, obstructive sleep apnea, hyperventilation syndrome, smoking or related illness, psychological factors, hormonal factors and drugs (NSAIDs, aspirin, beta blockers, ACE inhibitors) (Wechsler ME, 2014).

In severe asthma, inflammation can be dominated by eosinophils or neutrophils, or alternatively, both neutrophils and eosinophils act simultaneously, or neither. The number and distribution of inflammatory cells have been studied in saliva samples, bronchoalveolar lavage samples and samples taken from bronchial tubes. The most severe manifestations of asthma are associated with inflammation with both neutrophils and eosinophils.

In eosinophilic inflammation, the type 2 inflammatory response is central, where cytokines from Th2 helper cells (interleukin-4, -5 and -13) promote the secretion of immunoglobulin E (IgE) from plasma cells and e.g. eosinophil migration and activation. Eosinophils, on the other hand, secrete cytokines that promote inflammation and thereby respiratory tract dysfunction. The Th2 inflammatory response can be induced by, for example, an allergen, an infection or some external stimulus. Interleukin-5 (IL-5) is also an important mediator in the pathogenesis of severe eosinophilic asthma, which contributes to the differentiation, migration and activation of eosinophils. IL-5 is a cytokine secreted by at least lymphocytes and mast cells, but possibly also by eosinophils themselves. The mechanisms of neutrophilic inflammation in severe asthma are still poorly understood. However, in some patients with severe asthma, the airways no longer show signs of either of the above inflammatory processes, in which case the name "paucigranulocytic asthma" has been used. Even in this group, the mechanisms of severe asthma are still unclear and require further research. (Darveaux J, 2016, Israel E, 2017)

Biological drugs for severe asthma

The inflammatory mechanisms of severe asthma described above have been utilized in the development of new, targeted biological drugs. Currently in Finland, the IgE antibody omalizumab is used in severe allergic asthma and the IL-5 antibodies mepolizumab and reslizumab in severe eosinophilic asthma (Boyman O). Further studies are still needed on the benefits of biological drugs in the treatment of severe asthma, and more information and experience are needed especially in the selection of patients for biological drug treatment.

Omalizumab is a monoclonal IgE antibody that blocks the binding of IgE to its receptor on mast cells, dendritic cells, basophils, eosinophils and Langerhans cells. Omalizumab is the first monoclonal antibody approved for the treatment of severe allergic asthma. (Normansell R 2014). The clearest evidence has been seen in the reduction of exacerbations. Mepolizumab is a monoclonal IL-5 antibody whose effect in severe eosinophilic asthma is aimed at reducing eosinophilic inflammation. In studies, mepolizumab has been shown to reduce exacerbations in severe eosinophilic asthma, and it also seems to improve quality of life and reduce eosinophil levels in saliva and blood (Liu Y 2013). Reslizumab is a humanized IgG4-kappa IL-5 monoclonal antibody used in the treatment of severe eosinophilic asthma when other medications are inadequate. (Castro, M)

#### Aims of the study

1) The aim of the first part of the work was to find out whether asthma patients who received biological drug treatments for asthma have benefited from the medication in the form of a reduction in exacerbations, a reduction in the use of tablet cortisone or antimicrobial courses, a reduction in asthma symptoms or an improvement in the results of lung function tests.

2) The aim of the second part of the work is to find out the situation and treatment response of patients who have received biological drug treatments for asthma with regard to upper respiratory disease (chronic rhinosinusitis) and lung imaging findings (HRCT: atelectasis, bronchiectasis, bronchial thickening, nodules, mucus plugs, ground-glass changes, air blockage, reticulation (0 not at all, 1 on one side, 2 on both sides).

The information will be supplemented for those who have started new treatments and from others as needed: age, age, smoking (years of age), chronic/allergic rhinitis, osteoporosis, HRCT findings, BMI, OCS before biological treatments and the latest information, OCS courses during 12 months and the latest information, emergency room visits, antibiotic treatments, B-eos before and most recent, ACT before treatment and most recent, FEV1 (1, %, Z), FVC (1, %, Z), FEV1/FVC (1, %, Z), S-IgE, prick positivity (cat, dog, birch, timothy, dust mite, Aspergillus fumigatus), associated diseases (MCC, HTA, reflux, osteoporosis, COPD, fibrillation, sleep apnea, DM, hypothyroidism, depression, anxiety disorder), sputum bacterial, fungal and mycobacterial culture sample results (most recent if multiple taken, name of the microbe, +/++/+++). Information to be added: inhaled steroid (daily dose), po steroid (daily dose), LABA, LAMA, SABA, montelukast, theophylline (yes/no).

Regarding upper respiratory tract findings, the following are evaluated: NSO: fluid balance surfaces, mucosal edema, polyps; chronic rhinosinusitis 0 = no, 1 = yes (KNK or pulmonologist assessment), allergic rhinitis 0/1.

FESS, simple removal of polyps i.e. polypectomy, ethmoidectomy; antibiotic course(s) for sinusitis status: nasal polyposis (0/1) or wet in KNK status; nasal steroid yes/no, montelukast yes/no, po steroid continuously or in courses (dose); puncture culture findings (the most recent if several were taken, the name of the microbe, +/++/+++). In addition, biological drug treatment is recorded,

started (day), how long it was used (in months), appearance of upper respiratory tract symptoms after starting Biol drugs (worsened, unchanged, improved), whether polyps have recurred or worsened, whether upper respiratory tract procedures have been performed after starting biological drugs.

3) The goal of the third part of the work is to evaluate the effects of the digital asthma treatment path on asthma treatment results. The goal is to compare the number of exacerbations, symptoms, lung function test results and the need for medication in asthma patients treated according to the digital asthma treatment path with asthma patients who have not been treated with the treatment pa

#### 3. Plan

For the first part of the work, information was collected from the medical records of patients with severe asthma who received biological drug treatments in the HUS area since 2009. It was a retrospective study. In the second part of the work, information is sought on about 50 patients who have been treated with the digital path for asthma, and 50 patients who, at the same time, using a non-digital treatment path, have been treated in the allergy unit of the Skin and Allergy Hospital (HGD Study, HUH Goes Digital Study). Information to be searched is exacerbations, symptoms as assessed by the asthma symptom questionnaire, results of lung function tests and the need for medication. Based on the data, it is assessed whether there is a difference between the groups in treatment balance after 1 and 2 years of follow-up. The third part of the work currently utilizes the comprehensive asthma quality register of approx. 1,500 patients aged 18 or older and evaluates asthma treatment results, especially in the age group over 65 (n = 250), based on exacerbations, symptoms, lung function test results and the need for medication in a 2-year follow-up.